CLINICAL TRIAL: NCT05112055
Title: Microbiology and Treatment Outcome of Acute Exacerbation of Bronchiectasis in Hong Kong: a Prospective Study
Brief Title: Microbiology and Treatment Outcome of Acute Exacerbation of Bronchiectasis in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Wong Charles, Resident Specialist, Pamela Youde Nethersole Eastern Hospital
Other Study IDs: Pro_AEB_2021
Record Dates: First submitted 2021-10-08; First posted 2021-11-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchiectasis is a common disease worldwide with a high burden on healthcare resources. In Hong Kong (HK), local microbiological and clinical data regarding acute exacerbation of bronchiectasis (AEB) is lacking, in particular the frequency of pseudomonas aeruginosa (PA) in AEB is yet to be elucidated. A better understanding of the microbiology of AEB will provide evidence for judicious use of appropriate antibiotics in patients hospitalized for AEB to facilitate treatment and discharge.

This study aims to

1. elucidate the microbiology of AEB using both traditional culture and newer molecular multiplex methods,
2. identify factors associated with PA infection, and
3. describe the management and treatment outcome of AEB in HK

DETAILED DESCRIPTION:
Bronchiectasis is a common disease worldwide with a high burden on healthcare resources. In Hong Kong (HK), bronchiectasis ranked 5th highest as a cause of respiratory mortality, was the 6th highest reason for respiratory inpatient bed-days and was the 7th highest cause of respiratory hospitalization in Hong Kong in 2005.

Local microbiological and clinical data regarding acute exacerbation of bronchiectasis (AEB) is lacking, in particular the frequency of pseudomonas aeruginosa (PA) in AEB is yet to be elucidated. Traditional respiratory specimen takes time and lack sensitivity, a newer multiplex molecular method may be beneficial in improving sensitivity and reducing turnover time to detect pathogens involved in AEB. A better understanding of the microbiology of AEB will provide evidence for judicious use of appropriate antibiotics in patients hospitalized for AEB to facilitate treatment and discharge.

This study aims to

1. elucidate the microbiology of AEB using both traditional culture and newer molecular multiplex methods,
2. identify factors associated with PA infection, and
3. describe the management and treatment outcome of AEB in HK

ELIGIBILITY:
Inclusion Criteria

1. Patients admitted to participating hospital with a clinical diagnosis of acute exacerbation of bronchiectasis (AEB), defined as a change in bronchiectasis treatment associated with deterioration in three or more of the following key symptoms for at least 48 hours: cough; sputum volume and/or consistency; sputum purulence; breathlessness and/or exercise tolerance; fatigue and/or malaise; or haemoptysis.
2. Patients with an established diagnosis of bronchiectasis, defined as the presence of cough, shortness of breath, chronic sputum production, recurrent respiratory infection, or a combination thereof with CT thorax scan confirmation of the presence of bronchiectasis indicated by a bronchoarterial ratio of > 1, lack of tapering, airway visibility within 1 cm of the pleural surface, or a combination thereof.

Exclusion criteria

1. Patients unable to provide informed consent
2. Age < 18 years
3. Pregnancy
4. Bronchiectasis due to known cystic fibrosis
5. Bronchiectasis is not the main or co-dominant respiratory disease
6. Traction bronchiectasis due to interstitial lung disease
7. Prior lung transplantation for bronchiectasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients who are admitted to the participating hospital with acute exacerbations of bronchiectasis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbiology | 1 month
  Frequency of pseudomonas aeruginosa (PA) and non-PA infection
Risk factors for PA infection | 1 month
  Risk factors for PA infection

SECONDARY OUTCOMES:
Antibiotics use | 1 month
  Length of antibiotics use (days)
Length of stay | 1 month
  Length of hospital stay for AEB (days)
Recurrent exacerbation | 12 months
  Frequency of recurrent exacerbation
Mortality | 12 months
  Rate of all-cause mortality in 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Wong, Principal Investigator — Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Charles Wong, Hong Kong, Other, Hong Kong

IPD SHARING:
Plan to Share IPD: No